CLINICAL TRIAL: NCT00200122
Title: Restore Claims Characterization Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1617
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Refractory Pain Associated With Failed Back Surgery Syndrome, Epidural Fibrosis, Peripheral Causalgia, Complex Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation

SUMMARY:
The purpose of this study is to characterize the pain coverage capability of the RESTORE spinal cord stimulation (SCS) and assess health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Has chronic refractory pain associated with one of the conditions currently approved for spinal cord stimulation as follows: Failed Back Syndrome, Degenerative Disk Disease (DDD), Herniated Disk pain refractory to conservative and surgical interventions, Peripheral Causalgia, Complex Regional Pain Syndrome (CRPS) or Reflex Sympathetic Dystrophy (RSD).
* Primary pain in the lower half of the body.

Exclusion Criteria:

* Requires, or will in the future, diathermy treatments.
* Had implanted spinal cord stimulation system within the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to assesses the pain coverage capability of the RESTORE SCS system.

SECONDARY OUTCOMES:
Secondary outcome measures include pain relief, quality of life, function, patient and physician acceptance.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Contact Medtronic for Exact Location, Chicago, Illinois
  - Contact Medtronic for Exact Location, Indianapolis, Indiana
  - Contact Medtronic for Exact Location, Kansas City, Missouri
  - Contact Medtronic for Exact Location, Syosset, New York
  - Contact Medtronic for Exact Location, Eugene, Oregon
  - Contact Medtronic for Exact Location, Dallas, Texas
  - Contact Medtronic for Exact Location, San Antonio, Texas
  - Contact Medtronic for Exact Location, Huntington, West Virginia

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473